CLINICAL TRIAL: NCT02781883
Title: A Phase IIa, Open-label, Clinical Trial to Evaluate the Safety, Pharmacokinetics, Pharmacodynamics, and Efficacy of BP1001 (a Liposomal Grb2 Antisense Oligonucleotide) in Combination With Venetoclax Plus Decitabine in Patients With AML Who Are Ineligible for Intensive Induction Therapy
Brief Title: Clinical Trial of BP1001 in Combination With With Venetoclax Plus Decitabine in AML
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Bio-Path Holdings, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BP1001-201-AML
Record Dates: First submitted 2016-05-18; First posted 2016-05-25 (Estimated); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Acute Myeloid Leukemia (AML)
Keywords: Liposomal Grb-2 treatment of AML; Liposomal Grb-2 with Venetoclax plus decitabine for AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Untreated AML (Experimental): BP1001 in combination with Ventoclax plus decitabine
  Interventions: Drug: BP1001 in combination with Ventoclax plus decitabine
- Refractory/Relapsed AML (Experimental): BP1001 in combination with Ventoclax plus decitabine
  Interventions: Drug: BP1001 in combination with Ventoclax plus decitabine
- Refractory/Relapsed AML (ventoclax-intolerant or resistant) (Experimental): BP1001 + decitabine combination in patients who are resistant or intolerant of venetoclax-based treatment, or considered not optimal candidates for a venetoclax-based therapy.
  Interventions: Drug: BP1001 plus decitabine

INTERVENTIONS:
Drug: BP1001 in combination with Ventoclax plus decitabine — BP1001 in combination with Ventoclax plus decitabine
  Other Names: Liposomal Grb-2; L-Grb-2
  Arms: Refractory/Relapsed AML; Untreated AML
Drug: BP1001 plus decitabine — BP1001 plus decitabine in ventoclax intolerant or resistant subjects
  Other Names: Liposomal Grb-2; L-Grb-2
  Arms: Refractory/Relapsed AML (ventoclax-intolerant or resistant)

SUMMARY:
The primary objectives of this study are to assess: (1) whether the combination of BP1001 plus venetoclax plus decitabine provides greater efficacy (Complete Remission [CR], Complete Remission with incomplete hematologic recovery [CRi], Complete Remission with partial hematologic recovery [CRh], than venetoclax plus decitabine alone (by historical comparison) in participants with untreated AML that cannot or elect not to be treated with more intensive chemotherapy; (2) whether BP1001-based treatment provides greater efficacy (CR, CRi, CRh) than intensive chemotherapy (by historical comparison) in participants with refractory/relapsed AML.

DETAILED DESCRIPTION:
Improvement of clinical benefit in fragile AML patients while maintaining tolerability is an important area of further clinical development. Modern aggressive combination chemotherapy can induce CR in a significant proportion of patients with previously untreated AML, but relapse occurs in most unless patients undergo intensive allogeneic hematopoietic stem cell transplantation. Novel therapies are needed for these patients

The Grb2 gene has been mapped to the human chromosome region 17q22-qter, a region that is duplicated in leukemias and solid tumors, which may result in an increased copy number of the Grb2 gene product. As Grb2 is important for the transformation of murine hematopoietic cells, and the proliferation of human leukemia cells that express high levels of oncogenic tyrosine kinases, inhibition of Grb2 may have a significant impact on the natural history of leukemias. The study drug (BP1001) may be able to inhibit the cells from making Grb-2. Researchers hope that without this protein, the leukemia cells will die.

This represents an area in which targeted therapies might be of benefit to these patients. One such potential treatment is BP1001, liposomal anti-sense treatment directed against Growth Factor Receptor-Bound Protein 2 (Grb2). Decitabine is approved in Europe for the treatment of adult patients with newly diagnosed de novo or secondary acute myeloid leukemia (AML). In vitro studies in AML cells co-incubated with BP1001 and decitabine suggests that treatment of AML patients with decitabine followed by BP1001 may be a combination that could benefit patients with AML.

This Phase IIa, multicenter, study of BP1001 in combination with Ventoclax plus decitabine will enroll participants with AML who are not otherwise eligible for for intensive induction therapy.

This trial will utilize an open label design to assess the safety profile, PK, PD, and efficacy of of BP1001 in combination with Ventoclax plus decitabine to assess whether the combination of either provides greater efficacy than intensive chemotherapy alone.

There are 3 cohorts exploring three-drug combinations of BP1001, venetoclax and decitabine.

* Untreated AML patients will be treated with BP1001 plus venetoclax plus decitabine.
* Refractory/relapsed AML patients will also be treated with BP1001 plus venetoclax plus decitabine.
* A third cohort of BP1001 + decitabine is offered to refractory/relapsed AML patients who are venetoclax resistant or intolerant, or not considered by the investigator as optimal candidates for venetoclax-based therapy.

Each cohort will continue until approximately 19 evaluable participants have been investigated. At that point, enrollment will be placed on hold so that the Sponsor can perform an administrative review of the data to determine which treatment cohorts should continue with enrollment.

Should one or more cohorts continue with enrollment, the sample size will be increased up to 54 in the refractory/relapsed AML cohorts and 98 in the untreated AML cohort. These sample sizes for the study are based on the primary endpoint.

ELIGIBILITY:
Inclusion Criteria

At the time of Screening, participants must meet all of the following criteria to be considered eligible to participate in the study:

1. Adults ≥18 years of age
2. Females must be of non-childbearing potential, surgically sterile, postmenopausal, or practice adequate methods of contraception during the study and for 30 days after the last dose of study drug or decitabine
3. Males must agree to use an adequate method of contraception during the study and for at least 30 days after the last dose of study drug or decitabine
4. Histologically documented diagnosis (based on the 2008 World Health Organization [WHO] Classification) (Vardiman et al. 2009) of one of the following:

   1. Newly diagnosed untreated AML; or
   2. Untreated secondary AML, including AML that has progressed from MDS
   3. In some cases of AML associated with specific genetic abnormalities, however, the diagnosis of AML may be made if the blast count is less than 20% (Dohner et al. 2017) - specifically AML with t(15;17), t(8;21), inv(16), or t(16;16))
   4. Relapsed or Refractory AML
5. Investigator considers previously untreated participant ineligible for (or unwilling to receive) intensive induction therapy based on medical reasons, disease characteristics such as genetics, type of AML (untreated or secondary), or participant characteristics such as age, performance status, co-morbidities, organ dysfunctions, or patient election of low-intensity treatment
6. Eligible for venetoclax and decitabine therapy, based on Investigator assessment
7. Participant's WBC count is 25 x 10^9/L or less at study initiation. The use of leukapheresis or hydroxyurea before treatment initiation to achieve this is permitted.
8. Adequate hepatic and renal functions as defined by:

   1. Aspartate transaminase (AST) and alanine transaminase (ALT) ≤2.5 times the upper limit of normal (ULN); and
   2. Usually total bilirubin ≤ 1.5 ULN. In specific cases the PI may request a waiver of this requirement with medical justification and agreement with the medical monitor and Bio-Path holdings. And;
   3. Estimated glomerular filtration rate (eGFR) of at least 40 ml/min. These estimations can be calculated using any of the following methods (Appendix E: Formulas):

   i. Chronic Kidney Disease Epidemiology Collaboration (CKD-Epi) equation
   * GFR = 141 × min (Scr /κ, 1)^α × max(Scr /κ, 1)^-1.209 × 0.993^Age × 1.018 [if female] × 1.159 [if black] ii. Cockcroft gault equation
   * Cockcroft Gault equation utilizing the TBW (Total body weight) to calculate an estimated creatinine clearance
   * CrCl = [(140 - age) x TBW] / (Scr x 72) x 0.85 [if female] iii. Modification of Diet in Renal Disease (MDRD) Study equation
   * GFR (mL/min/1.73 m^2) = 175 × (Scr)^-1.154 × (Age)^-0.203 × 0.74 [if female] x 1.212 [if African American (AA)] iv. Creatinine clearance estimated by 24-hr urine collection for creatinine clearance
9. Documented Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
10. Recovered from the effects of any prior surgery, radiotherapy, or antineoplastic treatment (with the exception of alopecia), based on Investigator assessment
11. Willing and able to provide written informed consent 7.2. Exclusion Criteria

At the time of Screening, participants who meet any of the following criteria will be excluded from participating in the study:

1. Active non-hematologic or lymphoid malignancy other than AML treated with immuno- or chemotherapy within the previous 12 months except active non- melanoma, non-invasive skin cancer will be allowed.
2. Known, active leptomeningeal leukemia requiring intrathecal therapy. NOTE: Patients with a history of CNS disease may be allowed to participate based on at least 1 documented, negative spinal fluid assessment within 28 days prior to Screening
3. Isolated extramedullary leukemia without also meeting bone marrow criteria for acute leukemia (for AML usually = 20% blasts in BMA or BMB). Patients may have leukemia with lower blast counts (Dohner et al. 2010). Bio-Path Holdings and Investigator concurrence required.
4. Acute promyelocytic leukemia (APL) with t(15;17)(q22;q12) PML-RARA
5. Chronic myeloid leukemia (CML) in any phase
6. Receipt of any anti-cancer therapy within 14 days prior to C1D1, with the exception of hydroxyurea or anagrelide (within 24 hours), TKI (within 1day), a single dose of cytarabine (for proliferative disease)
7. Uncontrolled active, untreated, or progressive infection
8. Receipt of any investigational agent or study treatment within 30 days prior to C1D1
9. Females who are capable of becoming pregnant, test positive for pregnancy, or are breast-feeding during the Screening period, or intend to become pregnant or breast-feed during the course of the study or within 30 days after last dose of study drug
10. Serious intercurrent medical or psychiatric illness which, in the opinion of the Investigator, would interfere with the ability of the participant to complete the study
11. Known active or clinically significant hepatitis B infection (based on positive surface antigen [HBsAg]), hepatitis C infection (based on positive antibody [HCV Ab]), or human immunodeficiency virus (HIV-1 or HIV-2, based on positive antibody)
12. History of any hypersensitivity to venetoclax or decitabine, unless reaction is deemed irrelevant to the study by the Investigator and Medical Monitor
13. Presence of concurrent conditions that, in the opinion of the Investigator and/or Medical Monitor, may compromise the participant's ability to tolerate study treatment or interfere with any aspect of study conduct or interpretation of results. This includes but is not limited to, unstable or uncontrolled angina, New York Heart Association (NYHA) class III or IV congestive heart failure, uncontrolled and sustained hypertension, clinically significant cardiac dysrhythmia or clinically significant baseline ECG abnormality (e.g., QTcF >470 msec)
14. Within the past 6 months, has had any of the following: myocardial infarction, unstable angina pectoris, coronary/peripheral artery bypass graft, cerebrovascular accident or transient ischemic attack
15. Uncontrolled seizure disorder (i.e., seizures within the past 2 months)
16. Cannot receive live attenuated vaccine immunization prior to, during, or after treatment with venetoclax until B-cell recovery occurs
17. Unable or unwilling to communicate or cooperate with the Investigator or follow the protocol for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2016-05; Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Assessment of efficacy in untreated AML subjects by bone marrow aspirate or biopsy | 180 days
  Assess whether the combination of BP1001 and Ventoclax plus decitabine provides greater efficacy (Complete Remission [CR], Complete Remission with incomplete hematologic recovery [CRi], Complete Remission with partial hematologic recovery [CRh], than Ventoclax + decitabine alone (by historical comparison) with untreated AML that cannot or elect not to be treated with more intensive chemotherapy
Assessment of efficacy in refractory/relapsed AML subjects by bone marrow aspirate or biopsy | 180 days
  Assess whether BP1001-based treatment provides greater efficacy (CR, CRi, CRh) than intensive chemotherapy (by historical comparison) in participants with refractory/relapsed AML.

SECONDARY OUTCOMES:
Assessment of safety of BP1001 in combination with Ventoclax plus decitabine | 30 days
  Evaluate safety and toxicity of the combination of BP1001 with Ventoclax plus decitabine using non-hematologic and hematologic measures per NCI CTCAE criteria (with a safety run-in)
Assessment of the pharmacokinetics (PK) of BP1001 when given in combination with Ventoclax plus decitabine | 30 days
  Evaluate the in vivo PK using plasma to compute half life and elimination.
Assessment of Minimal Residual Disease (MRD) status in patients who achieve CR/CRi/CRh with BP1001-based treatment | 30 days
  Assess time to response from administration of BP1001-based treatment to CR, CRi, or CRh, negative MRD status as defined by the site and as available (Usually ≤ 0.1% by multi-parameter flow cytometry).
Assessment of Partial Remissions and blast count reductions. | 30 days
  Assessment of Partial Remissions (per Cheson, 2003), and blast count reductions (per Williams, 2016)
Assessment of overall survival | 180 days
  To assess event-free survival, overall survival, time to response, and duration of response from date of study entry to study closure or death.

CONTACTS AND LOCATIONS:
Overall Officials: Maro Ohanian, DO, Principal Investigator — M.D. Anderson Cancer Center
Locations (9):
- United States (9):
  - UCLA Medical Center, Los Angeles, California
  - Georgia Cancer Center at Augusta University, Augusta, Georgia
  - University of Kansas Cancer Center, Fairway, Kansas
  - New Jersey Hematology Oncology Associates, Brick, New Jersey
  - Laura & Isaac Pe lmutter Cancer Center at NYU Langone Health, New York, New York
  - Weill Cornell Medical College - New York - Presbyterian Hospital, New York, New York
  - University of Texas M.D. Anderson Cancer Center, Houston, Texas
  - Baylor Scott & White Research Institute, Temple, Texas
  - West Virginia University/Mary Babb Randolph Cancer Center, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No